CLINICAL TRIAL: NCT01550367
Title: Inhibiting the Systemic Autophagic Syndrome - A Phase I/II Study of Hydroxychloroquine and Aldesleukin in Renal Cell Carcinoma Patients (RCC). A Cytokine Working Group (CWG) Study
Brief Title: Study of Hydroxychloroquine and Aldesleukin in Renal Cell Carcinoma Patients (RCC)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Leonard Appleman (Other)
Collaborators: Prometheus Laboratories (Industry)
Responsible Party: Sponsor-Investigator, Leonard Appleman, MD, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCI 11-080
Record Dates: First submitted 2012-02-29; First posted 2012-03-12 (Estimated); Results first posted 2019-09-25 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Metastatic Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Hydroxychloroquine; Interleukin-2; aldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Hydroxychloroquine + IL-2 (Experimental): One course of treatment (84 days) will consist of high dose (600,000 IU/kg) bolus IL-2 administered intravenously every 8 hours on days 1-5 and 15-19 (maximum 14 doses/5 days of administration) and hydroxychloroquine (HCQ) orally started two weeks prior to IL-2 infusions and continued while able to take oral medication for up to 3 courses.
  Interventions: Drug: Hydroxychloroquine; Drug: IL-2

INTERVENTIONS:
Drug: Hydroxychloroquine — Continuous oral administration (at 600 mg/d) will be initiated prior to the first dose (day -14) given 14 days prior to initiation of the first dose of IL-2 and then daily or twice a day throughout all three treatment courses.
  Other Names: Plaquenil
Drug: IL-2 — 600,000 IU/kg IV bolus q 8 hrs x days 1-5 and 15-19 (maximum 28 doses - 14 per 5 day cycle) of each 84-day course
  Other Names: Aldesleukin

SUMMARY:
The main goal of the research study is to determine whether treating renal cell cancer patients with the study drug, hydroxychloroquine, along with IL-2, a standard treatment of kidney cancer that has spread to other parts of the body, can make the cancer easier to kill and eliminate. Another goal is to see how the study drug affects the body's immune cells which fight cancer cells.

DETAILED DESCRIPTION:
The rationale for combining the high dose bolus aldesleukin with hydroxychloroquine includes potential positive interactions on the immune regulatory side, non-overlapping toxicities, and potential for prolongation and increased number of responses based on murine studies conducted at the University of Pittsburgh. This study is a multi-center phase II study designed to estimate the efficacy of combination therapy of standard high dose bolus IL-2 and various doses of hydroxychloroquine therapy in metastatic RCC patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic renal cell carcinoma with predominantly clear cell histology.
* Have measurable disease by RECIST 1.1 criteria. For example, this would include tumor in the lung, liver, and retroperitoneum. Bone disease is difficult to follow and quantify and as a sole site would not be acceptable.
* Patients must be at least 4 weeks from radiation or surgery and recovered from all ill effects.
* Age ≥18 years.
* Karnofsky Performance Status ≥80%.
* Adequate end organ function:

  1. Hematologic: ANC ≥ 1000cells/uL, platelets ≥ 100,000/uL, hemoglobin ≥ 9g/dl (pre transfusion values used for prognostic factor, can be transfused or use recombinant erythropoietin growth factors but must not have active bleeding).
  2. Liver: AST ≤ 2 x ULN (upper limit of normal), serum total bilirubin ≤ 2 x ULN (except for patients with Gilbert's Syndrome).
  3. Renal: serum creatinine ≤ 1.5 mg/dL or estimated creatinine clearance ≥ 60ml/min using Cockcroft-Gault estimation using the formula per protocol.
  4. Pulmonary: FEV1 ≥ 2.0 liters or ≥ 75% of predicted for height and age. (PFTs are required for patients over 50 or with significant pulmonary or smoking history defined as >20 pack years or history of COPD/emphysema).
  5. Cardiac: No evidence of congestive heart failure, symptoms of coronary artery disease, myocardial infarction less than one year prior to entry, serious cardiac arrhythmias, or unstable angina. Patients who are over 40 or have had previous cardiac disease will be required to have a negative or low probability cardiac stress test for cardiac ischemia.
* Women should not be lactating and, if of childbearing age, have a negative pregnancy test within two weeks of entry to the study.
* Appropriate contraception in both genders.
* The patient must be competent and have signed informed consent.
* CNS: No history of cerebrovascular accident, transient ischemic attacks, central nervous system or brain metastases.

Exclusion Criteria:

* Patients who have previously received IL-2 are NOT eligible. Patients on HCQ in neoadjuvant protocols or in the past for clinical indications ARE eligible, as are patients who have previously received CTLA-4 and/or PD-1/PD-L1 antibodies.
* Concomitant second malignancy except for non-melanoma skin cancer, and non-invasive cancer such as cervical CIS, superficial bladder cancer without local recurrence or breast CIS.
* In patients with a prior history of invasive malignancy, less than five years in complete remission.
* Positive serology for HIV, hepatitis B or hepatitis C.
* Significant co-morbid illness such as uncontrolled diabetes or active infection that would preclude treatment on this regimen.
* Use of corticosteroids or other immunosuppression (if patient had been taking steroids, at least 2 weeks must have passed since the last dose).
* History of inflammatory bowel disease or other serious autoimmune disease. (Not including thyroiditis and rheumatoid arthritis). Patients already on hydroxychloroquine for such disorders are not eligible.
* Patients with organ allografts.
* Uncontrolled hypertension (BP >150/100 mmHg).
* Proteinuria dipstick > 3+ or ≥ 2gm/24 hours.
* Urine protein:creatinine ratio ≥ 1.0 at screening.
* Major surgery, open biopsy, significant traumatic injury within 28 days of starting treatment or anticipation of need for major surgical procedure during the course of the study.
* Minor surgical procedures, fine needle aspirations or core biopsies within 7 days prior to starting treatment. Central venous catheter placements are permitted.
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to starting treatment.
* Serious, non-healing wound, ulcer, or bone fracture.
* History of tumor-related or other serious hemorrhage, bleeding diathesis, or underlying coagulopathy.
* History of deep venous thrombosis, clinically significant peripheral vascular disease, or other thrombotic event.
* Inability to comply with study and/or follow-up procedures.
* Individuals with known history of glucose 6 phosphate deficiency are excluded from the trial (possible issue with HCQ tolerance).
* Patients with previously documented macular degeneration or diabetic retinopathy are excluded from the trial.
* Baseline EKG with QTc > 470 msec (including subjects on medication). Subjects with ventricular pacemaker for whom QT interval is not measurable will be eligible on a case-by-case basis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-03; Primary Completion 2018-02-06 (Actual); Study Completion 2019-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leonard J Appleman, MD, PhD, Principal Investigator — University of Pittsburgh
Locations (7):
- United States (7):
  - Loyola University Chicago, Maywood, Illinois
  - Indiana University Simon Cancer Center, Indianapolis, Indiana
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Dartmouth-Hitchcock Medical Center, Hanover, New Hampshire
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Providence Health & Services, Portland, Oregon
  - University of Pittsburgh Cancer Institute / UPMC CancerCenter, Pittsburgh, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Groups:
- Hydroxychloroquine (HCQ) (1,200 mg/d or 600 mg/d) + IL-2: One course of treatment (84 days) will consist of high dose (600,000 IU/kg) bolus IL-2 administered intravenously every 8 hours on days 1-5 and 15-19 (maximum 14 doses/5 days of administration) and hydroxychloroquine (HCQ) orally started two weeks prior to IL-2 infusions and continued while able to take oral medication for up to 3 courses.
  Hydroxychloroquine: Continuous oral administration (at 1,200 mg/d for initial (13) patients, then 600 mg/d for next (17) patients) was initiated prior to the first dose (day -14) given 14 days prior to initiation of the first dose of IL-2 and then daily or twice a day throughout all three treatment courses.
  IL-2: 600,000 IU/kg IV bolus q 8 hrs x days 1-5 and 15-19 (maximum 28 doses - 14 per 5 day cycle) of each 84-day course
  Note: Patients were initially treated at 1200 mg/d HCQ (13 patients), but after several unexpected adverse events, the dose of HCQ was reduced to 600 mg/d (17 patients).
Period: Overall Study
Arm/Group | Hydroxychloroquine (HCQ) (1,200 mg/d or 600 mg/d) + IL-2
Started | 30
1200 mg/d HCQ | 13
600 mg/d HCQ | 17
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Patients with metastatic RCC treated with IL-2 combined with hydroxychloroquine. Patients were initially treated at 1200 mg/d HCQ, but after several unexpected adverse events, dose was reduced to 600 mg/d.
Groups:
- Hydroxychloroquine (HCQ) (1,200 mg/d or 600 mg/d) + IL-2: One course of treatment (84 days) will consist of high dose (600,000 IU/kg) bolus IL-2 administered intravenously every 8 hours on days 1-5 and 15-19 (maximum 14 doses/5 days of administration) and hydroxychloroquine (HCQ) orally started two weeks prior to IL-2 infusions and continued while able to take oral medication for up to 3 courses.
  Hydroxychloroquine: Continuous oral administration (at 1,200 mg/d for initial (13) patients, then 600 mg/d for next (17) patients) was initiated prior to the first dose (day -14) given 14 days prior to initiation of the first dose of IL-2 and then daily or twice a day throughout all three treatment courses.
  IL-2: 600,000 IU/kg IV bolus q 8 hrs x days 1-5 and 15-19 (maximum 28 doses - 14 per 5 day cycle) of each 84-day course
  Note: Patients were initially treated at 1200 mg/d HCQ, but after several unexpected adverse events, the dose of HCQ was reduced to 600 mg/d.
Arm/Group | Hydroxychloroquine (HCQ) (1,200 mg/d or 600 mg/d) + IL-2
Number analyzed (Participants) | 30
Age, Continuous [Mean (Full Range); unit: years] — Population: Measure Analysis Population Description: Rows represent different dosage levels of HCQ.
  years
    1200 mg/d HCQ: number analyzed (Participants) | 13
    1200 mg/d HCQ | 58.2 [55.0 to 61.3]
    600 mg/d HCQ: number analyzed (Participants) | 17
    600 mg/d HCQ | 56.5 [52.0 to 60.9]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Rows represent different dosage levels of HCQ.
  Participants
    1200 mg/d HCQ: number analyzed (Participants) | 13
    1200 mg/d HCQ: Female | 4
    1200 mg/d HCQ: Male | 9
    600 mg/d HCQ: number analyzed (Participants) | 17
    600 mg/d HCQ: Female | 4
    600 mg/d HCQ: Male | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  All Patients: American Indian or Alaska Native | 0
  All Patients: Asian | 0
  All Patients: Native Hawaiian or Other Pacific Islander | 0
  All Patients: Black or African American | 0
  All Patients: White | 30
  All Patients: More than one race | 0
  All Patients: Unknown or Not Reported | 0
Karnofsky Performance Status (KPS) [Count of Participants; unit: Participants] — The Karnofsky Performance Status scores range from 0 to 100. A higher score means the patient is better able to carry out daily activities. Karnofsky Performance Status may be used to determine a patient's prognosis, to measure changes in a patient's ability to function, or to decide if a patient could be included in a clinical trial. Population: Indicating Karnofsky Status by HCQ dosage group
  Participants
    KPS Score - 1200 mg/d HCQ: number analyzed (Participants) | 13
    KPS Score - 1200 mg/d HCQ: KPS Score of 80 | 11
    KPS Score - 1200 mg/d HCQ: KPS Score of 90 | 1
    KPS Score - 1200 mg/d HCQ: KPS Score of 100 | 1
    KPS Score - 600 mg/d HCQ: number analyzed (Participants) | 17
    KPS Score - 600 mg/d HCQ: KPS Score of 80 | 13
    KPS Score - 600 mg/d HCQ: KPS Score of 90 | 0
    KPS Score - 600 mg/d HCQ: KPS Score of 100 | 4

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response - IL-2 Combined With Hydroxychloroquine (HCQ) at Either 1,200 mg/d or 600 mg/d) (All Patients)
Description: Clinical Response: per RECIST v1.1: Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (target or non-target) with reduction in short axis to <10 mm. Partial Response (PR): ≥30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study. Progressive Disease (PD):≥20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). The sum must also demonstrate an absolute increase of ≥5 mm. The appearance ≥1 new lesion(s) is considered progression.
Time Frame: Up to 3 years
Population: Patients with metastatic RCC treated with IL-2 combined with hydroxychloroquine (HCQ at either 1,200 mg/d or 600 mg/d) who were evaluable for clinical response. Note: Patients were initially treated at 1200 mg/d HCQ, but after several unexpected adverse events, dosing was reduced to 600 mg/d.
Measure: Count of Participants; unit: Participants
Groups:
- Hydroxychloroquine + IL-2: One course of treatment (84 days) will consist of high dose (600,000 IU/kg) bolus IL-2 administered intravenously every 8 hours on days 1-5 and 15-19 (maximum 14 doses/5 days of administration) and hydroxychloroquine (HCQ) orally started two weeks prior to IL-2 infusions and continued while able to take oral medication for up to 3 courses.
  Hydroxychloroquine: Continuous oral administration (at 600 mg/d) was initiated prior to the first dose (day -14) given 14 days prior to initiation of the first dose of IL-2 and then daily or twice a day throughout all three treatment courses.
  IL-2: 600,000 IU/kg IV bolus q 8 hrs x days 1-5 and 15-19 (maximum 28 doses - 14 per 5 day cycle) of each 84-day course
  Note: Patients were initially treated at 1200 mg/d HCQ, but after several unexpected adverse events, dose was reduced to 600 mg/d.
Arm/Group | Hydroxychloroquine + IL-2
Number analyzed (Participants) | 29
Participants
  Progressed Disease - All Patients | 9
  Stable Disease - All Patients | 14
  Partial Response - All Patients | 3
  Complete Response - All Patients | 3

2. Primary Outcome: Clinical Response - IL-2 Combined With Hydroxychloroquine (HCQ) at 1,200 mg/d
Description: as for outcome 1
Time Frame: Up to 3 years
Population: Patients with metastatic RCC treated with IL-2 combined with hydroxychloroquine (HCQ) 1,200 mg/d who were evaluable for clinical response.
Measure: Count of Participants; unit: Participants
Groups:
- Hydroxychloroquine + IL-2: One course of treatment (84 days) will consist of high dose (600,000 IU/kg) bolus IL-2 administered intravenously every 8 hours on days 1-5 and 15-19 (maximum 14 doses/5 days of administration) and hydroxychloroquine (HCQ) orally started two weeks prior to IL-2 infusions and continued while able to take oral medication for up to 3 courses.
  Hydroxychloroquine: Continuous oral administration (at 1,200 mg/d) will be initiated prior to the first dose (day -14) given 14 days prior to initiation of the first dose of IL-2 and then daily or twice a day throughout all three treatment courses.
Arm/Group | Hydroxychloroquine + IL-2
Number analyzed (Participants) | 12
Participants
  Progressed Disease | 5
  Stable Disease | 6
  Partial Response | 1
  Complete Response | 0

3. Primary Outcome: Clinical Response - IL-2 Combined With Hydroxychloroquine (HCQ) at 600 mg/d
Description: as for outcome 1
Time Frame: Up to 3 years
Population: Patients with metastatic RCC treated with IL-2 combined with hydroxychloroquine (HCQ) 600 mg/d who were evaluable for clinical response.
Measure: Count of Participants; unit: Participants
Groups:
- Hydroxychloroquine + IL-2: One course of treatment (84 days) will consist of high dose (600,000 IU/kg) bolus IL-2 administered intravenously every 8 hours on days 1-5 and 15-19 (maximum 14 doses/5 days of administration) and hydroxychloroquine (HCQ) orally started two weeks prior to IL-2 infusions and continued while able to take oral medication for up to 3 courses.
  Hydroxychloroquine: Continuous oral administration (at 600 mg/d) was initiated prior to the first dose (day -14) given 14 days prior to initiation of the first dose of IL-2 and then daily or twice a day throughout all three treatment courses.
Arm/Group | Hydroxychloroquine + IL-2
Number analyzed (Participants) | 17
Participants
  Progressed Disease | 4
  Stable Disease | 8
  Partial Response | 2
  Complete Response | 3

4. Secondary Outcome: Overall Survival (OS)
Description: Time from date of first protocol treatment until the date of death, or censored at date of last contact.
Time Frame: Up to 3 years
Population: Patients with metastatic RCC treated with IL-2 combined with hydroxychloroquine (HCQ).
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Hydroxychloroquine (HCQ) (1,200 mg/d or 600 mg/d) + IL-2: One course of treatment (84 days) consisted of high dose (600,000 IU/kg) bolus IL-2 administered intravenously every 8 hours on days 1-5 and 15-19 (maximum 14 doses/5 days of administration) and hydroxychloroquine (HCQ) orally started two weeks prior to IL-2 infusions and continued while able to take oral medication for up to 3 courses.
  Hydroxychloroquine: Continuous oral administration (at 1,200 mg/d for initial (13) patients, then 600 mg/d for next (17) patients) was initiated prior to the first dose (day -14) given 14 days prior to initiation of the first dose of IL-2 and then daily or twice a day throughout all three treatment courses.
  IL-2: 600,000 IU/kg IV bolus q 8 hrs x days 1-5 and 15-19 (maximum 28 doses - 14 per 5 day cycle) of each 84-day course
  Note: Patients were initially treated at 1200 mg/d HCQ, but after several unexpected adverse events, the dose of HCQ was reduced to 600 mg/d.
Arm/Group | Hydroxychloroquine (HCQ) (1,200 mg/d or 600 mg/d) + IL-2
Number analyzed (Participants) | 30
months | NA [29.6 to NA] — Median and upper limit estimated overall survival in this trial is not yet achieved due to insufficient number of events (deaths).

5. Secondary Outcome: Progression-free Survival (PFS)
Description: Time from the date of first protocol treatment until the date disease progression criteria are met (in responding patients progression criteria uses the reference of the smallest measurements recorded since the treatment started) or is censored at date of last disease assessment for those who have not progressed. Per RECIST 1.1, Progressive Disease (PD) is defined as ≥20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). The sum must also demonstrate an absolute increase of ≥5 mm. The appearance ≥1 new lesion(s) is considered progression.
Time Frame: Up to 3 years
Population: Patients with metastatic RCC treated with IL-2 combined with hydroxychloroquine (HCQ) at either 600 mg/d or 1,200 mg/d.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Hydroxychloroquine (HCQ) (1,200 mg/d or 600 mg/d) + IL-2
Number analyzed (Participants) | 30
months | 5.5 [3.0 to 14.0]

6. Secondary Outcome: Number of Doses of IL-2 + HCQ
Description: Number of doses of IL-2 administered during the first course of therapy.
Time Frame: Up to 3 years
Population: Patients that received at least one dose of study treatment (IL-2 + either 1,200 HCQ or 600 mg/d HCQ).
Measure: Mean (95% Confidence Interval); unit: doses
Arm/Group | Hydroxychloroquine (HCQ) (1,200 mg/d or 600 mg/d) + IL-2
Number analyzed (Participants) | 30
doses
  1200 mg/d HCQ: number analyzed (Participants) | 13
  1200 mg/d HCQ | 12.8 [9.8 to 15.7]
  600 mg/d HCQ: number analyzed (Participants) | 17
  600 mg/d HCQ | 13.2 [11.0 to 15.4]

7. Secondary Outcome: Frequency of Grade III and Grade IV Toxicities
Description: Number of specified categories of grade III and IV or unexpected or rare toxicities occurring during the first course (up until the end of cycle 1) of IL-2 treatment.
Time Frame: Up to 3 years
Population: Patients that received at least one dose (cycle) of study treatment (IL-2 + either 1,200 HCQ or 600 mg/d HCQ) and experienced specified categories of toxicities.
Measure: Number; unit: events
Arm/Group | Hydroxychloroquine (HCQ) (1,200 mg/d or 600 mg/d) + IL-2
Number analyzed (Participants) | 30
events
  Hypotension | 5
  Gastrointestinal | 1
  Hematologic | 1
  Pulmonary | 1
  Renal/electrolytes | 4
  Psychiatric | 3

8. Secondary Outcome: Worst Grade of Adverse Event Experienced
Description: Number of participants who experienced Grade 2-5 adverse events.
Time Frame: Up to 3 years
Population: Patients that received at least one dose of study treatment (IL-2 + either 1,200 HCQ or 600 mg/d HCQ).
Measure: Count of Participants; unit: Participants
Arm/Group | Hydroxychloroquine (HCQ) (1,200 mg/d or 600 mg/d) + IL-2
Number analyzed (Participants) | 30
Participants
  1200 mg/d HCQ: number analyzed (Participants) | 13
  1200 mg/d HCQ: Grade 2 adverse event | 1
  1200 mg/d HCQ: Grade 3 adverse event | 4
  1200 mg/d HCQ: Grade 4 adverse event | 7
  1200 mg/d HCQ: Grade 5 adverse event | 1
  600 mg/d HCQ: number analyzed (Participants) | 17
  600 mg/d HCQ: Grade 2 adverse event | 0
  600 mg/d HCQ: Grade 3 adverse event | 4
  600 mg/d HCQ: Grade 4 adverse event | 13
  600 mg/d HCQ: Grade 5 adverse event | 0

9. Secondary Outcome: Worst Grade of Adverse Event At Least Possibly Related to Treatment Experienced
Description: Number of participants who experienced Grade 2-5 adverse events that were at least possibly related to study treatment.
Time Frame: Up to 3 years
Population: Patients that received at least one dose of study treatment (IL-2 + either 1,200 HCQ or 600 mg/d HCQ).
Measure: Count of Participants; unit: Participants
Groups:
- Hydroxychloroquine (HCQ) (1,200 mg/d or 600 mg/d) + IL-2: One course of treatment (84 days) consisted of high dose (600,000 IU/kg) bolus IL-2 administered intravenously every 8 hours on days 1-5 and 15-19 (maximum 14 doses/5 days of administration) and hydroxychloroquine (HCQ) orally started two weeks prior to IL-2 infusions and continued while able to take oral medication for up to 3 courses.
  Hydroxychloroquine: Continuous oral administration (at 1,200 mg/d for initial (13) patients, then 600 mg/d for next (17) patients) was initiated prior to the first dose (day -14) given 14 days prior to initiation of the first dose of IL-2 and then daily or twice a day throughout all three treatment courses.
  IL-2: 600,000 IU/kg IV bolus q 8 hrs x days 1-5 and 15-19 (maximum 28 doses - 14 per 5 day cycle) of each 84-day course
  Note: Patients were initially treated at 1200 mg/d HCQ (13 patients), but after several unexpected adverse events, the dose of HCQ was reduced to 600 mg/d (17 patients).
Arm/Group | Hydroxychloroquine (HCQ) (1,200 mg/d or 600 mg/d) + IL-2
Number analyzed (Participants) | 30
Participants
  1200 mg/d HCQ: number analyzed (Participants) | 13
  1200 mg/d HCQ: Grade 2 adverse event | 1
  1200 mg/d HCQ: Grade 3 adverse event | 5
  1200 mg/d HCQ: Grade 4 adverse event | 7
  600 mg/d HCQ: number analyzed (Participants) | 17
  600 mg/d HCQ: Grade 2 adverse event | 0
  600 mg/d HCQ: Grade 3 adverse event | 4
  600 mg/d HCQ: Grade 4 adverse event | 13

10. Secondary Outcome: Worst Grade of Adverse Event At Least Probably Related to Treatment Experienced
Description: Number of participants who experienced Grade 2-5 adverse events that were at least probably related to study treatment.
Time Frame: Up to 3 years
Population: Patients that received at least one dose of study treatment (IL-2 + either 1,200 HCQ or 600 mg/d HCQ).
Measure: Count of Participants; unit: Participants
Arm/Group | Hydroxychloroquine (HCQ) (1,200 mg/d or 600 mg/d) + IL-2
Number analyzed (Participants) | 30
Participants
  1200 mg/d HCQ: number analyzed (Participants) | 13
  1200 mg/d HCQ: Grade 2 adverse event | 1
  1200 mg/d HCQ: Grade 3 adverse event | 5
  1200 mg/d HCQ: Grade 4 adverse event | 7
  600 mg/d HCQ: number analyzed (Participants) | 17
  600 mg/d HCQ: Grade 2 adverse event | 2
  600 mg/d HCQ: Grade 3 adverse event | 4
  600 mg/d HCQ: Grade 4 adverse event | 11

11. Secondary Outcome: Serum Lactate Dehydrogenase
Description: Number of participants with either high serum lactate dehydrogenase (> 1.5 times upper limit of normal) or normal lactate dehydrogenase.
Time Frame: Up to 2 years
Population: Patients that received study treatment for whom LDH was able to be measured from clinical samples and determined to be either normal or high.
Measure: Count of Participants; unit: Participants
Arm/Group | Hydroxychloroquine (HCQ) (1,200 mg/d or 600 mg/d) + IL-2
Number analyzed (Participants) | 30
Participants
  Normal LDH: number analyzed (Participants) | 28
  Normal LDH: 1200 mg/d HCQ | 11
  Normal LDH: 600 mg/d HCQ | 17
  High LDH: number analyzed (Participants) | 2
  High LDH: 1200 mg/d HCQ | 2
  High LDH: 600 mg/d HCQ | 0

12. Secondary Outcome: Hemoglobin Levels
Description: Low hemoglobin levels (less than the lower limit of normal (13.2 g/dL)) are considered to be unfavorable.
Time Frame: Up to 3 years
Population: Patient that received study treatment for whom hemoglobin levels were able to be measured from clinical samples and determined to be either normal or low.
Measure: Count of Participants; unit: Participants
Arm/Group | Hydroxychloroquine (HCQ) (1,200 mg/d or 600 mg/d) + IL-2
Number analyzed (Participants) | 30
Participants
  Low hemoglobin level: number analyzed (Participants) | 9
  Low hemoglobin level: 1200 mg/d HCQ | 6
  Low hemoglobin level: 600 mg/d HCQ | 3
  Normal hemoglobin level: number analyzed (Participants) | 21
  Normal hemoglobin level: 1200 mg/d HCQ | 7
  Normal hemoglobin level: 600 mg/d HCQ | 14

13. Secondary Outcome: Serum Calcium Levels (Corrected)
Description: Number of patients with either normal or high serum calcium levels. High serum calcium levels are considered to be clinically unfavorable.
Time Frame: Up to 3 years
Population: Patients that received study treatment for whom serum calcium levels were able to be measured from clinical samples and determined to be either normal or high.
Measure: Count of Participants; unit: Participants
Arm/Group | Hydroxychloroquine (HCQ) (1,200 mg/d or 600 mg/d) + IL-2
Number analyzed (Participants) | 30
Participants
  Normal Calcium: number analyzed (Participants) | 27
  Normal Calcium: 1200 mg/d HCQ | 13
  Normal Calcium: 600 mg/d HCQ | 14
  High Calcium: number analyzed (Participants) | 3
  High Calcium: 1200 mg/d HCQ | 0
  High Calcium: 600 mg/d HCQ | 3

14. Secondary Outcome: Prior Nephrectomy
Description: Number of patients with history of a prior nephrectomy (surgical removal of a kidney) or no history of a prior nephrectomy.
Time Frame: Up to 3 years
Population: Patients that received study treatment, with or without a history of nephrectomy (surgical removal of a kidney).
Measure: Count of Participants; unit: Participants
Arm/Group | Hydroxychloroquine (HCQ) (1,200 mg/d or 600 mg/d) + IL-2
Number analyzed (Participants) | 30
Participants
  No Prior Nephrectomy: number analyzed (Participants) | 3
  No Prior Nephrectomy: 600 mg/d HCQ | 3
  No Prior Nephrectomy: 1200 mg/d HCQ | 0
  Prior Nephrectomy: number analyzed (Participants) | 27
  Prior Nephrectomy: 600 mg/d HCQ | 14
  Prior Nephrectomy: 1200 mg/d HCQ | 13

15. Secondary Outcome: Number of Participants With Low Karnofsky Performance Status
Description: Karnofsky performance status is a standard way of measuring the ability of cancer patients to perform ordinary tasks. The Karnofsky Performance Status scores range from 0 to 100. A higher score means the patient is better able to carry out daily activities. Karnofsky Performance Status may be used to determine a patient's prognosis, to measure changes in a patient's ability to function, or to decide if a patient should be included in the trial. A low Karnofsky performance status (<80%) is considered to be unfavorable.
Time Frame: Up to 3 years
Population: Patient that received study treatment for whom Karnofsky performance status was able to be assessed.
Measure: Count of Participants; unit: Participants
Arm/Group | Hydroxychloroquine (HCQ) (1,200 mg/d or 600 mg/d) + IL-2
Number analyzed (Participants) | 30
Participants
  1200 mg/d HCQ: number analyzed (Participants) | 13
  1200 mg/d HCQ | 0
  600 mg/d HCQ: number analyzed (Participants) | 17
  600 mg/d HCQ | 0

16. Secondary Outcome: Natural Killer (NK) Cells
Description: Percentage of Natural Killer (NK) cells per ml of blood. NK cells are lymphocytes with the ability to kill tumor cells without deliberate immunization or activation.
Time Frame: Up to 3 years
Population: Patients that received study treatment for whom Natural Killer (NK) cells were able to be measured.
Measure: Mean (Full Range); unit: percentage of cells
Arm/Group | Hydroxychloroquine (HCQ) (1,200 mg/d or 600 mg/d) + IL-2
Number analyzed (Participants) | 30
percentage of cells | 38.4 [3.7 to 67.3]

17. Secondary Outcome: Myeloid Derived Suppressor Cell (MDSC)
Description: Percentage of Myeloid Derived Suppressor Cell per ml of blood. MDSC immune cells originate from bone marrow stem cells and strongly expand in cancer.
Time Frame: Up to 3 years
Population: Patients that received study treatment for whom MDSC were able to be measured.
Measure: Mean (Full Range); unit: percentage of cells/mL
Arm/Group | Hydroxychloroquine (HCQ) (1,200 mg/d or 600 mg/d) + IL-2
Number analyzed (Participants) | 30
percentage of cells/mL | 11.3 [4.4 to 23.6]

18. Secondary Outcome: Regulatory T Cells (Treg)
Description: Percentage of Regulatory T cells per ml of blood. High levels of Tregs in the tumor microenvironment are associated with poor prognosis in many cancers by suppressing the body's anti-tumor immune response.
Time Frame: Up to 3 years
Population: Patients that received study treatment for whom Regulatory T cells (Treg) were able to be measured.
Measure: Mean (Full Range); unit: percentage of cells/mL
Arm/Group | Hydroxychloroquine (HCQ) (1,200 mg/d or 600 mg/d) + IL-2
Number analyzed (Participants) | 30
percentage of cells/mL | 10.5 [1.7 to 20.8]

19. Secondary Outcome: Plasmacytoid Dendritic Cells (pDC)
Description: Percentage of Plasmacytoid dendritic cells per ml of blood. In cancer, pDC are malignant immune cells that demonstrate an impaired response that can contribute to the establishment of an immunosuppressive tumor microenvironment.
Time Frame: Up to 3 years
Population: Patients that received study treatment for whom Plasmacytoid dendritic Cells (pDC) were able to be measured.
Measure: Mean (Full Range); unit: percentage of cells/mL
Arm/Group | Hydroxychloroquine (HCQ) (1,200 mg/d or 600 mg/d) + IL-2
Number analyzed (Participants) | 30
percentage of cells/mL | 0.3 [0.1 to 0.8]

20. Secondary Outcome: T-cell Lymphocytes
Description: Percentage of T-cell lymphocytes in blood as cells per ml. T-cells are a subtype of white blood cells which play a key role in the immune system and fighting cancer.
Time Frame: Up to 3 years
Population: Patients that received study treatment for whom T-Cells were able to be measured.
Measure: Mean (Full Range); unit: percentage of cells/mL
Arm/Group | Hydroxychloroquine (HCQ) (1,200 mg/d or 600 mg/d) + IL-2
Number analyzed (Participants) | 30
percentage of cells/mL | 63.9 [17.7 to 80.5]

21. Secondary Outcome: Conventional Dendritic Cells (cDC)
Description: Percentage of Conventional Dendritic Cells (cDC) per ml of blood. cDC reside in tissues and once activated, migrate to draining lymph nodes to promote adaptive immune responses.
Time Frame: Up to 3 years
Population: Patients that received study treatment for whom Conventional Dendritic Cells (cDC) were able to be measured.
Measure: Mean (Full Range); unit: percentage of cells/mL
Arm/Group | Hydroxychloroquine (HCQ) (1,200 mg/d or 600 mg/d) + IL-2
Number analyzed (Participants) | 30
percentage of cells/mL | 0.6 [0 to 1.5]

ADVERSE EVENTS:
Time Frame: Up to 3 years for cohort.
Groups:
- Hydroxychloroquine (HCQ) (1,200 mg/d ) + IL-2: One course of treatment (84 days) will consist of high dose (600,000 IU/kg) bolus IL-2 administered intravenously every 8 hours on days 1-5 and 15-19 (maximum 14 doses/5 days of administration) and hydroxychloroquine (HCQ) orally started two weeks prior to IL-2 infusions and continued while able to take oral medication for up to 3 courses.
  Hydroxychloroquine: Continuous oral administration (at 1,200 mg/d (initial (13) patients) was initiated prior to the first dose (day -14) given 14 days prior to initiation of the first dose of IL-2 and then daily or twice a day throughout all three treatment courses.
  IL-2: 600,000 IU/kg IV bolus q 8 hrs x days 1-5 and 15-19 (maximum 28 doses - 14 per 5 day cycle) of each 84-day course
  Note: Patients were initially treated at 1200 mg/d HCQ (13 patients), but after several unexpected adverse events, the dose of HCQ was reduced to 600 mg/d (17 patients).
- Hydroxychloroquine (HCQ) (600 mg/d) + IL-2: One course of treatment (84 days) will consist of high dose (600,000 IU/kg) bolus IL-2 administered intravenously every 8 hours on days 1-5 and 15-19 (maximum 14 doses/5 days of administration) and hydroxychloroquine (HCQ) orally started two weeks prior to IL-2 infusions and continued while able to take oral medication for up to 3 courses.
  Hydroxychloroquine: Continuous oral administration at 600 mg/d (17 patients) was initiated prior to the first dose (day -14) given 14 days prior to initiation of the first dose of IL-2 and then daily or twice a day throughout all three treatment courses.
  IL-2: 600,000 IU/kg IV bolus q 8 hrs x days 1-5 and 15-19 (maximum 28 doses - 14 per 5 day cycle) of each 84-day course
  Note: Patients were initially treated at 1200 mg/d HCQ (13 patients), but after several unexpected adverse events, the dose of HCQ was reduced to 600 mg/d (17 patients).
Arm/Group | Hydroxychloroquine (HCQ) (1,200 mg/d ) + IL-2 | Hydroxychloroquine (HCQ) (600 mg/d) + IL-2
All-Cause Mortality (participants affected / at risk) | 9/13 | 2/17
Serious Adverse Events (participants affected / at risk) | 12/13 | 17/17
Other Adverse Events (participants affected / at risk) | 13/13 | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydroxychloroquine (HCQ) (1,200 mg/d ) + IL-2 (N=13) | Hydroxychloroquine (HCQ) (600 mg/d) + IL-2 (N=17)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Akathisia (Nervous system disorders) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 2 (4)
Anxiety (Psychiatric disorders) | 1 (2) | 2 (2)
Apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 2 (2) | 1 (1)
Cardiac disorders - Other, specify (Cardiac disorders) | 2 (2) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0)
Death NOS (General disorders) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 (8) | 3 (6)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2) | 2 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 6 (19) | 15 (41)
Hypotension (Vascular disorders) | 6 (9) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Investigations - Other, specify (Investigations) | 0 (0) | 1 (2)
Lipase increased (Investigations) | 2 (8) | 1 (1)
Lymphocyte count decreased (Investigations) | 6 (37) | 13 (66)
Mucositis oral (Gastrointestinal disorders) | 1 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 2 (2)
Platelet count decreased (Investigations) | 3 (4) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 2 (2) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Serum amylase increased (Investigations) | 3 (4) | 0 (0)
Urinary retention (Renal and urinary disorders) | 5 (10) | 3 (6)
Urine output decreased (Investigations) | 1 (1) | 0 (0)
White blood cell decreased (Investigations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydroxychloroquine (HCQ) (1,200 mg/d ) + IL-2 (N=13) | Hydroxychloroquine (HCQ) (600 mg/d) + IL-2 (N=17)
Abdominal pain (Gastrointestinal disorders) | 3 (6) | 3 (3)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 3 (3) | 0 (0)
Agitation (Psychiatric disorders) | 2 (2) | 1 (1)
Akathisia (Nervous system disorders) | 1 (2) | 2 (2)
Alanine aminotransferase increased (Investigations) | 6 (9) | 8 (12)
Alkaline phosphatase increased (Investigations) | 8 (26) | 6 (16)
Allergic reaction (Immune system disorders) | 0 (0) | 3 (3)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 8 (41) | 13 (50)
Anorexia (Metabolism and nutrition disorders) | 6 (11) | 6 (13)
Anxiety (Psychiatric disorders) | 5 (14) | 11 (17)
Apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (2) | 2 (2)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 7 (10) | 8 (9)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Bile duct stenosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 8 (23) | 9 (22)
Blurred vision (Eye disorders) | 0 (0) | 1 (1)
CPK increased (Investigations) | 3 (5) | 1 (1)
Capillary leak syndrome (Vascular disorders) | 0 (0) | 4 (4)
Cardiac disorders - Other, specify (Cardiac disorders) | 4 (6) | 5 (10)
Cardiac troponin I increased (Investigations) | 1 (1) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 9 (16) | 8 (17)
Confusion (Psychiatric disorders) | 3 (4) | 2 (2)
Constipation (Gastrointestinal disorders) | 4 (4) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (5) | 7 (7)
Creatinine increased (Investigations) | 7 (39) | 12 (64)
Death NOS (General disorders) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 11 (27) | 13 (28)
Dizziness (Nervous system disorders) | 1 (1) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 2 (3) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 7 (10) | 9 (20)
Dysgeusia (Nervous system disorders) | 3 (4) | 3 (6)
Dyspepsia (Gastrointestinal disorders) | 3 (5) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 10 (15) | 7 (8)
Edema face (General disorders) | 0 (0) | 2 (2)
Edema limbs (General disorders) | 9 (19) | 10 (18)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Eye disorders - Other, specify (Eye disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fatigue (General disorders) | 9 (28) | 12 (34)
Fever (General disorders) | 3 (4) | 7 (23)
Flashing lights (Eye disorders) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 8 (15) | 8 (19)
Gait disturbance (General disorders) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 2 (2) | 2 (3)
General disorders and administration site conditions - Other, specify (General disorders) | 8 (18) | 9 (18)
Hallucinations (Psychiatric disorders) | 1 (1) | 4 (4)
Headache (Nervous system disorders) | 4 (4) | 4 (5)
Heart failure (Cardiac disorders) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 2 (2) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hot flashes (Vascular disorders) | 0 (0) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (2) | 2 (5)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 4 (4)
Hyperkalemia (Metabolism and nutrition disorders) | 6 (13) | 4 (10)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1) | 3 (6)
Hypertension (Vascular disorders) | 1 (1) | 4 (6)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 8 (61) | 14 (77)
Hypocalcemia (Metabolism and nutrition disorders) | 7 (14) | 12 (30)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 3 (3) | 6 (9)
Hypomagnesemia (Metabolism and nutrition disorders) | 11 (28) | 16 (48)
Hyponatremia (Metabolism and nutrition disorders) | 9 (28) | 13 (36)
Hypophosphatemia (Metabolism and nutrition disorders) | 10 (37) | 16 (75)
Hypotension (Vascular disorders) | 11 (26) | 12 (29)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
INR increased (Investigations) | 0 (0) | 4 (5)
Insomnia (Psychiatric disorders) | 5 (6) | 5 (5)
Investigations - Other, specify (Investigations) | 5 (9) | 11 (15)
Lipase increased (Investigations) | 4 (21) | 6 (12)
Localized edema (General disorders) | 0 (0) | 1 (2)
Lymphocyte count decreased (Investigations) | 6 (43) | 13 (76)
Malaise (General disorders) | 3 (3) | 0 (0)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 2 (4) | 1 (1)
Mucosal infection (Infections and infestations) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 6 (10) | 7 (11)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 2 (3) | 2 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 12 (30) | 14 (40)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Nervous system disorders - Other, specify (Nervous system disorders) | 3 (3) | 3 (6)
Neutrophil count decreased (Investigations) | 2 (3) | 4 (6)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (2) | 0 (0)
Pain (General disorders) | 1 (1) | 5 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Pancreatitis (Gastrointestinal disorders) | 3 (4) | 0 (0)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 1 (1)
Photophobia (Eye disorders) | 1 (1) | 1 (1)
Platelet count decreased (Investigations) | 8 (25) | 12 (45)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 6 (8) | 4 (11)
Pruritus (Skin and subcutaneous tissue disorders) | 11 (22) | 10 (21)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 2 (2) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (5)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 2 (2) | 4 (5)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 5 (8)
Restlessness (Psychiatric disorders) | 0 (0) | 1 (1)
Serum amylase increased (Investigations) | 4 (18) | 2 (7)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 7 (14) | 6 (8)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 3 (3) | 4 (4)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1)
Superficial thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 2 (2)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 1 (3)
Urinary retention (Renal and urinary disorders) | 6 (12) | 5 (10)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2)
Urine output decreased (Investigations) | 1 (1) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Vascular disorders - Other, specify (Vascular disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 9 (21) | 11 (25)
Weight gain (Investigations) | 5 (6) | 8 (12)
Weight loss (Investigations) | 2 (3) | 3 (4)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
White blood cell decreased (Investigations) | 5 (8) | 6 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-05): https://cdn.clinicaltrials.gov/large-docs/67/NCT01550367/Prot_SAP_000.pdf